CLINICAL TRIAL: NCT00683982
Title: Nitazoxanide vs Probiotics in the Treatment of Acute Rotavirus Diarrhea in Children: A Randomized Single Blind Controlled Trial in Bolivian Children
Brief Title: Use of Nitazoxanide and Probiotics in Acute Diarrhea Secondary to Rotavirus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Pediatrico Albina de Patino (Other)
Responsible Party: Carlos Teran Escalera/Jefe de Comite de Investigacion, Centro Pediatrico Albina Patiño
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROT261179; PROT261179B
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2008-05-26 (Estimated); Status verified 2008-05

CONDITIONS: Diarrhea; Rotavirus Infection
Keywords: nitazoxanide; Probiotics; Diarrhea; Rotavirus; Children
MeSH Terms: conditions — Diarrhea; Rotavirus Infections | interventions — nitazoxanide; Probiotics

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): This group will receive oral nitazoxanide preparation
  Interventions: Drug: Nitazoxanide
- 2 (Active Comparator): This group will receive a mix combination of probiotics
  Interventions: Drug: Probiotic mix preparation
- 3 (Placebo Comparator): This is the control group receiving only oral or systemic hydration solutions
  Interventions: Other: Oral hydration solutions

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide 15mg/Kg/day twice day for 3 days
  Other Names: Noxom; Givotan
  Arms: 1
Drug: Probiotic mix preparation — Probiotic preparation 1 gram twice a day for 5 days
  Other Names: Probiotic
  Arms: 2
Other: Oral hydration solutions — Oral hydration solutions as needed
  Other Names: Rehsal 60; 2.5% Glucosaline
  Arms: 3

SUMMARY:
Nitazoxanide has proved an cytoprotective effect against rotavirus infection. How it could be clinically important in time of hospitalization and reduction of duration of diarrhea secondary to rotavirus?

DETAILED DESCRIPTION:
Nitazoxanide has demonstrated a cytoprotective effect against rotavirus, reducing duration time of diarrhea in comparison to placebo in previous studies. In the current study, based in those results, we design a randomized single-blind controlled trial, in order to asses the effectiveness of nitazoxanide and probiotics in comparison with a control group

ELIGIBILITY:
Inclusion Criteria:

* Positive stool sample for rotavirus test

Exclusion Criteria:

* Severe malnourishment
* Severe dehydration
* History of diarrhea more than 3 days previous hospitalization
* Use of antibiotics, probiotics or nitazoxanide 3 weeks before admission
* Systemic infections
* Severe chronic disease
* Mixed enteric infections besides rotavirus

Ages: 28 Days to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2007-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea | Hours

SECONDARY OUTCOMES:
Duration of hospitalization | hours

CONTACTS AND LOCATIONS:
Overall Officials: Carlos N Teran, M.D, Study Director — Centro Pediatrico Albina Patiño
Locations (1):
- Centro Pediatrico Albina Patiño, Cochabamba, Departamento de Cochabamba, Bolivia